CLINICAL TRIAL: NCT01528072
Title: Post Market Surveillance for the Dynesys Spinal System, Assessing Safety and Fusion.
Brief Title: Dynesys Spinal System Post Market 522 Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated at request of FDA
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMU2010-10S
Record Dates: First submitted 2012-02-02; First posted 2012-02-07 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Degenerative Spondylolisthesis; Pseudoarthrosis
Keywords: Dynesys Dynamic Stabilization System; Spondylolithesis; pseudoarthrosis; neurologic impairment; failed fusion
MeSH Terms: conditions — Pseudarthrosis; Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dynesys System (Experimental): All patients will receive the Dynesys System and all patients will be compared to historical literature control. Dynesys Spinal System will be used for all subjects.
  Interventions: Device: Dynesys Spinal System

INTERVENTIONS:
Device: Dynesys Spinal System — Dynesys Spinal System will be used for all subjects

SUMMARY:
The purpose of this study is to assess the safety and fusion rates following posterior lateral fusion with the Dynesys Spinal System used as an adjunct to fusion and compare to literature control.

DETAILED DESCRIPTION:
Study is meant to assess the safety and fusion rates following posterior lateral fusion with the Dynesys Spinal System.

ELIGIBILITY:
Inclusion Criteria:

1. Skeletally mature between the ages of 20-80
2. Candidate for posterior lateral fusion between T1-S1 with autograft
3. Degenerative spondylolisthesis with evidence of neurologic impairment or failed previous fusion (pseudoarthrosis)
4. Symptoms of leg and/or back pain
5. Non-responsive to conservative/non-surgical treatment for at least three (3) months
6. Must be willing and able to comply with study requirements; including complete necessary study paperwork and return for required follow-up visits

Exclusion Criteria:

1. Active systemic or local infection
2. Obesity
3. Use of interbody device
4. Pregnancy
5. Mental illness
6. Incarceration
7. Alcohol or drug abuse
8. Severe osteoporosis or osteopenia
9. Use in the cervical spine
10. Sensitivities/allergy to metals, polymers, polyethylene, polycarbonate urethane and polyethylene terephthalate
11. Soft tissue deficit not allowing sound closure
12. Any medical or physical condition that would preclude the potential benefit of spinal implant surgery
13. Congenital abnormalities, tumors or other conditions that would prevent secure component fixation that has the potential to decrease the useful life of the device
14. Active malignancy or other significant medical comorbidities
15. Any medical or mental condition which would put the patient at high risk due to the severity of surgery
16. Inadequate pedicles of the thoracic, lumbar and sacral vertebrae
17. Patient unwilling or unable to follow postoperative instructions

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2012-03; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Batts, Study Director — Zimmer Biomet Spine
Locations (9):
- United States (9):
  - Neurological Surgery of Southern Ill, Belleville, Illinois
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Pine Heights Medical Center, Baltimore, Maryland
  - NYU - Center for Musculoskeletal Care, New York, New York
  - Riverhills Healthcare, Inc, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - OrthopaediCare, Willow Grove, Pennsylvania
  - Danville Orthopedics and Spine, Danville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the time between signing consent and application of treatment 13 subjects were discontinued. Out of 153 enrolled there were: 5- screen failures; 1- withdraw consent; 5- insurance denials; 2- Removed by investigator.
Groups:
- Dynesys System: Dynesys Spinal System will be used for all subjects
Period: Overall Study
Arm/Group | Dynesys System
Started | 140
Completed | 66
Not Completed | 74
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 1
Not completed — Determined not eligible by AEAC | 1
Not completed — Missed Visit | 2
Not completed — Lost to Follow-up | 5
Not completed — Explanted | 2
Not completed — Site Closure | 4
Not completed — Death | 2
Not completed — Early Termination of Study | 52

BASELINE CHARACTERISTICS:
Population: Baseline variables were summarized for all subjects who were eligible, enrolled in the study and underwent a surgical procedure where the Dynesys® Spinal System was implanted.
Arm/Group | Dynesys System
Number analyzed (Participants) | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88
  Male | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: inches] | 65.7 (3.7)
Weight [Mean (Standard Deviation); unit: pounds] | 184.6 (39.6)
BMI [Mean (Standard Deviation); unit: (kg/mg^2)] | 30 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Fusion Rates
Description: Fusion was defined by meeting three criteria:
  * rotation < 5° between motion segments on flexion-extension radiographs
  * translation < 3 mm between motion segments on flexion-extension radiographs
  * presence of bridging bone. Fusion assessment for each patient was categorized as one of the four defined outcomes: fused, not fused, partial fusion, or UA (unable to assess). Efficacy was confirmed by the achievement of fusion in the experimental group when compared to the rate established in a literature control.
Time Frame: 24 months post surgery date
Population: Sixty-six (66) out of the original 140 implanted subjects completed their 24 month follow up. Sixty-one (61) subjects completed 24month radiograph for analysis of the primary end point.
Measure: Count of Participants; unit: Participants
Arm/Group | Dynesys System
Number analyzed (Participants) | 61
Participants
  Proportion fused | 33
  Proportion not fused | 19
  Proportion with Partial Fusion | 5
  Proportion unable to assess | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of surgery through the participants last visit; up to 48months.
Description: Any unfavorable and unintended sign, symptom, or disease associated with the use of an investigational product, whether or not related to the investigational product, taking into consideration the patient history, surgical history, histological analysis as well as explants evaluation. Events may be complications, observations (including radiographic), change in patient condition or related/unrelated death. A change indicating worsening as reported on an assessment is an adverse event.
Arm/Group | Dynesys System
All-Cause Mortality (participants affected / at risk) | 2/139
Serious Adverse Events (participants affected / at risk) | 33/139
Other Adverse Events (participants affected / at risk) | 71/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dynesys System (N=139)
Acidosis (Metabolism and nutrition disorders) | 1 (1) — Diabetic Ketoacidosis
Allergic reaction (Immune system disorders) | 1 (1) — Reaction to Tramadol
Anemia (Blood and lymphatic system disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) — Clostridium difficile
Fever (General disorders) | 1 (1)
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Other- Iliac artery aneurysm (Vascular disorders) | 1 (2)
Intracranial hemorrhage (Nervous system disorders) | 2 (2)
Meningitis (Infections and infestations) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Other- Adjacent level disease (Musculoskeletal and connective tissue disorders) | 4 (4) — Lumbar
Other- Bilateral knee arthroplasty (Surgical and medical procedures) | 1 (1)
Other- Mucinous adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Other- Postoperative pneumonia (Infections and infestations) | 1 (1)
Other- Spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) — Lumbar
Other- Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) — Cervical
Other- Total hip arthoroplasty (Musculoskeletal and connective tissue disorders) | 2 (2)
Other- Urinary hesitancy (Renal and urinary disorders) | 1 (1)
Other- Wound (Injury, poisoning and procedural complications) | 1 (1) — Leg
Pseudomeningocele (Nervous system disorders) | 1 (1)
Radiculitis (Nervous system disorders) | 5 (5)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) — Cellulitis
Superficial thrombophlebitis (Vascular disorders) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Visceral arterial ischemia (Vascular disorders) | 1 (1) — Ischemic bowel
Other- Incision site necrosis (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dynesys System (N=139)
Ileus (Gastrointestinal disorders) | 2 (2)
Wound infection (Infections and infestations) | 2 (2)
Intraoperative neurological injury (Injury, poisoning and procedural complications) | 5 (5) — Dural tear
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) — Leg
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) — Knee
Buttock pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) — Hip
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) — Ankle
Neuralgia (Nervous system disorders) | 5 (5) — Leg
Neuralgia (Nervous system disorders) | 2 (2) — Neck
Paresthesia (Nervous system disorders) | 4 (4) — Leg
Radiculitis (Nervous system disorders) | 3 (3)
Hypotension (Vascular disorders) | 2 (2)
Other- Adjacent level disease (Nervous system disorders) | 3 (3)
Other- Pain in leg (Nervous system disorders) | 2 (2)
Other- Pain low back (Nervous system disorders) | 4 (4)
Other- pain in back (Nervous system disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Early termination lead to a significant subset of subjects to not make it to the final follow up time interval. This resulted in small numbers of subjects analyzed for fusion and literature control was not used as planned originally in protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2011-12-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT01528072/Prot_SAP_ICF_000.pdf